CLINICAL TRIAL: NCT06822920
Title: Monitoring the Use of Collagen Dura Membrane in the Post-market Phase
Brief Title: Post-Market Clinical Investigation Plan - Collagen Dura Membranes (DM & DMO)
Acronym: DM&DMO
Status: Recruiting | Type: Observational
Sponsor: Collagen Matrix (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP.010
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Repair of Dura Mater

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Monitoring the Use of Collagen Dura Membrane in the Post-market phase

DETAILED DESCRIPTION:
A multi-center clinical series of 110 patients treated with Collagen Dura Substitute Membrane (DuraMatrix & DuraMatrix Onlay) for a dural defect in the dura mater will be evaluated prospectively. Patients will have follow-up time points through at least 6-9 months which align with the lifetime of the device. The primary endpoint of the study will be the presence of adverse events leakage that require surgical intervention, will be evaluated at each follow-up time point. The secondary endpoint of the study will be adverse events i.e. infection, Cerebrospinal fluid leak (CSF) and Pseudomeningocele. No patient records or personal identifying information will be disclosed to Collagen Matrix.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a dural defect requiring repair with a dural substitute.

Exclusion Criteria:

* There are no subject restrictions for the study other than patients with known allergy to bovine collagen products as specified in the contraindications of the Instructions for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject device is intended for all patient populations. The following population is excluded from the study:-
  * Pregnant Women
  * Subjects requiring Legally Authorized Representative
  * Subjects under 18 years of age
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of the occurrence of adverse event requiring surgical intervention | 6-9 months

SECONDARY OUTCOMES:
Adverse events i.e., infection, CSF leak and Pseudomeningocele | 6-9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Collagen of Wisconsin, Milwaukee, Wisconsin, United States